CLINICAL TRIAL: NCT01830972
Title: An Open-label Phase 2 Extension Study to Evaluate the Long Term Safety and Efficacy of Sialic Acid-Extended Release (SA-ER) Tablets and Sialic Acid-Immediate Release (SA-IR) Capsules in Patients With GNE Myopathy or Hereditary Inclusion Body Myopathy
Brief Title: An Open Label Phase 2 Extension Study of Higher Dose Sialic Acid-Extended Release (SA-ER) Tablets and Sialic Acid-Immediate Release (SA-IR) Capsules in Patients With Glucosamine (UDP-N-acetyl)-2-Epimerase (GNE) Myopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UX001-CL202
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: GNE Myopathy; Hereditary Inclusion Body Myopathy (HIBM)
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crossover Participants (Experimental): Participants completing the 48-week study (UX001-CL201; NCT01517880) were enrolled into Part I of the study:
  * Part I: participants continued on 6 g/day SA-ER for 12 weeks
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment 4 times per day [QID]) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
  Interventions: Drug: SA-ER 500 mg; Drug: SA-IR 500 mg
- Naïve Participants (Experimental): Treatment naïve participants with GNE myopathy were enrolled into Part II of the study:
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment QID) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
  Interventions: Drug: SA-ER 500 mg; Drug: SA-IR 500 mg

INTERVENTIONS:
Drug: SA-ER 500 mg — oral tablets
Drug: SA-IR 500 mg — oral capsules

SUMMARY:
The safety objectives of the study are to: evaluate additional long-term safety of SA-ER treatment of participants with GNE myopathy previously treated with SA-ER at dose of 6g/day (Part I); evaluate the safety of 12g /day SA (delivered by 1.5g of SA-ER tablets and 1.5g of SA-IR capsules 4 times per day) in the treatment of participants with GNE myopathy (Part II) over a 6 month treatment period; evaluate the safety of SA treatment at both 6g/day and 12 g/day (Part III [SA-ER/SA-IR] and Part IV [SA-ER]).

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in, and successful completion of the UX001-CL201 (NCT01517880) protocol OR (for 10 treatment naïve subjects):

  * Have a confirmed diagnosis of GNE Myopathy
  * Aged 18 -65 years of age, inclusive
  * Able to walk ≥ 200 meters and < 80% of predicted normal during the 6-Minute Walk Test (6MWT; orthotics and assistive devices allowed)
* Must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Must be willing and able to comply with all study procedures
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study
* Females of childbearing potential must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause for at least two years, or have had tubal ligation at least one year prior to Baseline, or who have had total hysterectomy

Exclusion Criteria:

* Use of any investigational product (other than SA-ER tablets) to treat GNE myopathy
* Ingestion of N-acetyl-D-mannosamine (ManNAc) or similar SA-producing compounds
* Pregnant or breastfeeding at Baseline or planning to become pregnant (self or partner) at any time during the study
* Has had any hypersensitivity to SA or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* Have any co-morbid conditions, including unstable major organ-system disease(s) that in the opinion of the investigator, places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-06-04 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Medical Center, New York, New York
- Hadassah University Hospital, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completing study UX001-CL201 (NCT01517880) were eligible to continue treatment under this protocol. Additional participants with glucosamine (UDP-N-acetyl)-2-epimerase (GNE) myopathy were enrolled to assess Sialic Acid Extended Release/Sialic Acid Immediate Release (SA-ER/SA-IR) in a treatment naïve population.
Pre-assignment Details: A total of 46 crossover participants started the study in Part 1, with an additional 13 naive participants starting the study in Part 2.
Groups:
- Crossover Participants: Participants completing the 48-week study (UX001-CL201) were enrolled into Part I of the study:
  * Part I: participants continued on 6 g/day SA-ER for approximately 6 months
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment 4 times per day [QID]) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
Period: Part I
Arm/Group | Crossover Participants | Naïve Participants
Started | 46 | 0 (Not applicable; participants in this arm entered during Part 2.)
Completed | 46 | 0 (Not applicable; participants in this arm entered during Part 2.)
Not Completed | 0 | 0
Period: Part II
Arm/Group | Crossover Participants | Naïve Participants
Started | 46 | 13 (Entered study at Part 2)
Completed | 44 | 11
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Part III
Arm/Group | Crossover Participants | Naïve Participants
Started | 44 (2 participants withdrew consent and did not enter Part 3) | 11
Completed | 42 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Noncompliance | 1 | 0
Period: Part IV
Arm/Group | Crossover Participants | Naïve Participants
Started | 42 | 11
Completed | 39 | 10
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Non-Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline at the start of Part II (upon study entry for Naïve Participants) is presented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Participants | Naïve Participants | Total
Number analyzed (Participants) | 46 | 13 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.55) | 35.6 (10.97) | 39.9 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 8 | 37
  Male | 17 | 5 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 13 | 51
  Asian | 8 | 0 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic/Latino | 44 | 13 | 57
  Hispanic/Latino | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An adverse event (AE) is defined as any untoward medical occurrence, whether or not considered drug related. A serious AE (SAE) is an AE that at any dose results in any of the following: death, a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect. TEAEs include all adverse events that start on or after the first dose of study medication, or adverse events that are present prior to the first dose of study medication, but their severity or relationship increases after the first dose of study medication up to and including 30 days after the final study medication dosing date. TEAEs were graded as mild (grade 1), moderate (grade 2), severe (grade 3), life-threatening (grade 4), or death (grade 5). TEAE relationship to study medication was classified as not related, possibly related, or probably related.
Time Frame: From first dose of study drug until up to 30 days after the last dose of study drug. Mean (SD) duration of treatment was 1170.0 (170.2) days for Crossover Participants and 897 (380) days for Naïve Participants
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Participants; 6 g/Day; Crossover Participants: 12 g/Day; Crossover Participants: Any Dose: Participants completing the 48-week study (UX001-CL201) were enrolled into Part I of the study:
  * Part I: participants continued on 6 g/day SA-ER for approximately 6 months
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment 4 times per day [QID]) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
- Naïve Participants: 6 g/Day; Naïve Participants: 12 g/Day: Treatment naïve participants with GNE myopathy were enrolled into Part II of the study:
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment QID) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
- Overall: Any Dose: Participants completing the 48-week study (UX001-CL201) were enrolled into Part I of the study and treatment naïve participants with GNE myopathy were enrolled into Part II of the study:
  * Part I: participants continued on 6 g/day SA-ER for approximately 6 months
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment 4 times per day [QID]) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
Arm/Group | Crossover Participants; 6 g/Day | Crossover Participants: 12 g/Day | Crossover Participants: Any Dose | Naïve Participants: 6 g/Day | Naïve Participants: 12 g/Day | Overall: Any Dose
Number analyzed (Participants) | 46 | 46 | 46 | 1 | 13 | 59
Participants
  >/= 1 TEAE | 43 | 46 | 46 | 1 | 13 | 59
  TEAE Maximum Severity = Grade 1 | 19 | 23 | 15 | 0 | 5 | 20
  TEAE Maximum Severity = Grade 2 | 22 | 23 | 29 | 1 | 7 | 36
  TEAE Maximum Severity = Grade 3 | 2 | 0 | 2 | 0 | 1 | 3
  TEAE Maximum Severity = Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE Maximum Severity = Grade 5 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment Related TEAEs | 26 | 40 | 45 | 1 | 11 | 56
  Serious TEAEs | 2 | 0 | 2 | 0 | 1 | 3
  TEAEs Causing Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Clinically Significant Changes From Baseline in Vital Signs, Physical and Neurological Examination Findings and Laboratory Evaluations
Time Frame: as for outcome 1
Population: Clinically significant changes from Baseline for vital signs, physical and neurological examination findings and laboratory evaluations were recorded as AEs and are reported as part of the Safety section of this record and Outcome Measure 1.
Arm/Group | Crossover Participants | Naïve Participants
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Interval History: Has the Participant Experienced Any New Conditions or Exacerbations of an Existing Condition Since Last Study Visit?
Description: Each interval history was intended to record any signs, symptoms, or events (e.g., falls, changes in medications or therapies) experienced by the participant since the prior study visit that were not related to study procedure(s) performed at prior study visits or study drug. Interval history may have included exacerbation or improvement in existing medical conditions (including the clinical manifestations of GNE myopathy) that might have interfered with study participation, safety, and/or positively or negatively impact performance of functional assessments.
Time Frame: Part I: Baseline (Study UX001-CL201 Week 48), Month 6; Part II-IV: Baseline, Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 33, 36, study termination
Population: All participants who received at least one dose of study drug. Participant "n" at each time point includes those with a yes or no response. Naïve Participants did not enter the study until Part II.
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Participants | Naïve Participants
Number analyzed (Participants) | 46 | 13
Participants
  Part I Baseline (Study UX001-CL201 Week 48): Yes: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): Yes | 29 |
  Part I Baseline (Study UX001-CL201 Week 48): No: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): No | 17 |
  Part I Month 6: Yes: number analyzed (Participants) | 6 | 0
  Part I Month 6: Yes | 6 |
  Part I Month 6: No: number analyzed (Participants) | 6 | 0
  Part I Month 6: No | 0 |
  Part II-IV Baseline: Yes: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: Yes | 28 | 0
  Part II-IV Baseline: No: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: No | 18 | 1
  Part II-IV Month 1: Yes | 36 | 12
  Part II-IV Month 1: No | 10 | 1
  Part II-IV Month 3: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: Yes | 0 | 1
  Part II-IV Month 3: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: No | 0 | 0
  Part II-IV Month 6: Yes: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: Yes | 27 | 7
  Part II-IV Month 6: No: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: No | 19 | 4
  Part II-IV Month 9: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: Yes | 0 | 1
  Part II-IV Month 9: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: No | 0 | 0
  Part II-IV Month 12: Yes: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: Yes | 29 | 6
  Part II-IV Month 12: No: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: No | 17 | 4
  Part II-IV Month 15: Yes: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: Yes | 4 | 5
  Part II-IV Month 15: No: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: No | 1 | 3
  Part II-IV Month 18: Yes: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: Yes | 18 | 3
  Part II-IV Month 18: No: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: No | 21 | 0
  Part II-IV Month 21: Yes: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: Yes | 18 | 8
  Part II-IV Month 21: No: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: No | 12 | 3
  Part II-IV Month 24: Yes: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: Yes | 12 | 0
  Part II-IV Month 24: No: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: No | 2 | 0
  Part II-IV Month 27: Yes: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: Yes | 21 | 5
  Part II-IV Month 27: No: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: No | 21 | 5
  Part II-IV Month 33: Yes: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: Yes | 11 | 2
  Part II-IV Month 33: No: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: No | 5 | 1
  Part II-IV Month 36: Yes: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: Yes | 10 | 6
  Part II-IV Month 36: No: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: No | 13 | 1
  Part II-IV Termination: Yes: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: Yes | 0 | 0
  Part II-IV Termination: No: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: No | 1 | 0

4. Primary Outcome: Interval History: Has the Participant Started Taking Any New Medications or Discontinued Any Medications Since the Study Visit?
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Participants | Naïve Participants
Number analyzed (Participants) | 46 | 13
Participants
  Part I Baseline (Study UX001-CL201 Week 48): Yes: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): Yes | 21 |
  Part I Baseline (Study UX001-CL201 Week 48): No: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): No | 25 |
  Part I Month 6: Yes: number analyzed (Participants) | 6 | 0
  Part I Month 6: Yes | 4 |
  Part I Month 6: No: number analyzed (Participants) | 6 | 0
  Part I Month 6: No | 2 |
  Part II-IV Baseline: Yes: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: Yes | 23 | 0
  Part II-IV Baseline: No: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: No | 23 | 1
  Part II-IV Month 1: Yes | 15 | 4
  Part II-IV Month 1: No | 31 | 9
  Part II-IV Month 3: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: Yes | 0 | 1
  Part II-IV Month 3: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: No | 0 | 0
  Part II-IV Month 6: Yes: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: Yes | 24 | 7
  Part II-IV Month 6: No: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: No | 22 | 4
  Part II-IV Month 9: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: Yes | 0 | 1
  Part II-IV Month 9: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: No | 0 | 0
  Part II-IV Month 12: Yes: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: Yes | 27 | 5
  Part II-IV Month 12: No: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: No | 19 | 5
  Part II-IV Month 15: Yes: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: Yes | 4 | 3
  Part II-IV Month 15: No: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: No | 1 | 5
  Part II-IV Month 18: Yes: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: Yes | 17 | 2
  Part II-IV Month 18: No: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: No | 22 | 1
  Part II-IV Month 21: Yes: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: Yes | 19 | 7
  Part II-IV Month 21: No: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: No | 11 | 4
  Part II-IV Month 24: Yes: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: Yes | 10 | 0
  Part II-IV Month 24: No: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: No | 4 | 0
  Part II-IV Month 27: Yes: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: Yes | 19 | 6
  Part II-IV Month 27: No: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: No | 23 | 4
  Part II-IV Month 33: Yes: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: Yes | 12 | 2
  Part II-IV Month 33: No: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: No | 4 | 1
  Part II-IV Month 36: Yes: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: Yes | 12 | 5
  Part II-IV Month 36: No: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: No | 11 | 2
  Part II-IV Termination: Yes: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: Yes | 0 | 0
  Part II-IV Termination: No: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: No | 1 | 0

5. Primary Outcome: Interval History: Has the Participant Started Receiving Any New Therapy or Discontinued Any Therapies Since Last Study Visit?
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Participants | Naïve Participants
Number analyzed (Participants) | 46 | 13
Participants
  Part I Baseline (Study UX001-CL201 Week 48): Yes: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): Yes | 5 |
  Part I Baseline (Study UX001-CL201 Week 48): No: number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48): No | 41 |
  Part I Month 6: Yes: number analyzed (Participants) | 6 | 0
  Part I Month 6: Yes | 3 |
  Part I Month 6: No: number analyzed (Participants) | 6 | 0
  Part I Month 6: No | 3 |
  Part II-IV Baseline: Yes: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: Yes | 9 | 0
  Part II-IV Baseline: No: number analyzed (Participants) | 46 | 1
  Part II-IV Baseline: No | 37 | 1
  Part II-IV Month 1: Yes | 4 | 0
  Part II-IV Month 1: No | 42 | 13
  Part II-IV Month 3: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: Yes | 0 | 0
  Part II-IV Month 3: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 3: No | 0 | 1
  Part II-IV Month 6: Yes: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: Yes | 9 | 4
  Part II-IV Month 6: No: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6: No | 37 | 7
  Part II-IV Month 9: Yes: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: Yes | 0 | 0
  Part II-IV Month 9: No: number analyzed (Participants) | 0 | 1
  Part II-IV Month 9: No | 0 | 1
  Part II-IV Month 12: Yes: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: Yes | 5 | 2
  Part II-IV Month 12: No: number analyzed (Participants) | 46 | 10
  Part II-IV Month 12: No | 41 | 8
  Part II-IV Month 15: Yes: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: Yes | 0 | 0
  Part II-IV Month 15: No: number analyzed (Participants) | 5 | 8
  Part II-IV Month 15: No | 5 | 8
  Part II-IV Month 18: Yes: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: Yes | 4 | 0
  Part II-IV Month 18: No: number analyzed (Participants) | 39 | 3
  Part II-IV Month 18: No | 35 | 3
  Part II-IV Month 21: Yes: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: Yes | 3 | 0
  Part II-IV Month 21: No: number analyzed (Participants) | 30 | 11
  Part II-IV Month 21: No | 27 | 11
  Part II-IV Month 24: Yes: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: Yes | 2 | 0
  Part II-IV Month 24: No: number analyzed (Participants) | 14 | 0
  Part II-IV Month 24: No | 12 | 0
  Part II-IV Month 27: Yes: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: Yes | 4 | 1
  Part II-IV Month 27: No: number analyzed (Participants) | 42 | 10
  Part II-IV Month 27: No | 38 | 9
  Part II-IV Month 33: Yes: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: Yes | 3 | 0
  Part II-IV Month 33: No: number analyzed (Participants) | 16 | 3
  Part II-IV Month 33: No | 13 | 3
  Part II-IV Month 36: Yes: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: Yes | 3 | 3
  Part II-IV Month 36: No: number analyzed (Participants) | 23 | 7
  Part II-IV Month 36: No | 20 | 4
  Part II-IV Termination: Yes: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: Yes | 0 | 0
  Part II-IV Termination: No: number analyzed (Participants) | 1 | 0
  Part II-IV Termination: No | 1 | 0

6. Primary Outcome: Interval History: Typical Number of Falls Per Year
Description: as for outcome 3
Time Frame: Part I: Baseline (Study UX001-CL201 Week 48), Month 6; Part II-IV: Baseline, Months 1, 6, 12, 18, 24, 30, 36, study termination
Population: All participants who received at least one dose of study drug. Naïve Participants did not enter the study until Part II.
Measure: Mean (Standard Deviation); unit: falls
Arm/Group | Crossover Participants | Naïve Participants
Number analyzed (Participants) | 46 | 13
falls
  Part I Baseline (Study UX001-CL201 Week 48): number analyzed (Participants) | 46 | 0
  Part I Baseline (Study UX001-CL201 Week 48) | 11.0 (53.63) |
  Part I Month 6: number analyzed (Participants) | 6 | 0
  Part I Month 6 | 3.8 (3.54) |
  Part II-IV Baseline | 14.1 (53.66) | 6.0 (6.19)
  Part II-IV Month 1: number analyzed (Participants) | 46 | 12
  Part II-IV Month 1 | 6.8 (9.60) | 7.3 (6.31)
  Part II-IV Month 6: number analyzed (Participants) | 46 | 11
  Part II-IV Month 6 | 8.0 (11.87) | 5.6 (6.39)
  Part II-IV Month 12: number analyzed (Participants) | 46 | 11
  Part II-IV Month 12 | 5.4 (8.94) | 5.1 (3.51)
  Part II-IV Month 18: number analyzed (Participants) | 44 | 11
  Part II-IV Month 18 | 7.8 (14.58) | 6.0 (4.15)
  Part II-IV Month 24: number analyzed (Participants) | 43 | 11
  Part II-IV Month 24 | 9.4 (28.23) | 4.5 (3.05)
  Part II-IV Month 30: number analyzed (Participants) | 41 | 11
  Part II-IV Month 30 | 6.2 (10.03) | 5.0 (6.56)
  Part II-IV Month 36: number analyzed (Participants) | 39 | 10
  Part II-IV Month 36 | 5.4 (9.03) | 7.6 (10.88)
  Part II-IV Termination: number analyzed (Participants) | 1 | 1
  Part II-IV Termination | 4.0 (NA) — SD is not applicable for 1 participant. | 12.0 (NA) — SD is not applicable for 1 participant.

ADVERSE EVENTS:
Time Frame: From first dose of study drug until up to 30 days after the last dose of study drug. Mean (SD) duration of treatment was 1170.0 (170.2) days for Crossover Participants and 897 (380) days for Naive Participants.
Description: TEAEs are presented. TEAEs include all adverse events that start on or after the first dose of study medication, or adverse events that are present prior to the first dose of study medication, but their severity or relationship increases after the first dose of study medication up to and including 30 days after the final study medication dosing date.
Groups:
- Crossover Participants; 6 g/Day; Crossover Participants: 12 g/Day; Crossover Participants: Any Dose: Participants completing the 48-week study (UX001-CL201) were enrolled into Part I of the study:
  * Part I: participants continued on 6 g/day SA-ER for approximately 6 months
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment QID) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
- Overall: Any Dose: Participants completing the 48-week study (UX001-CL201) were enrolled into Part I of the study and treatment naïve participants with GNE myopathy were enrolled into Part II of the study:
  * Part I: participants continued on 6 g/day SA-ER for approximately 6 months
  * Part II: 12 g/day SA (1.5 g of SA-ER and 1.5 g of SA-IR treatment QID) for 36 months
  * Part III: 6 g/day or 12 g/day SA (both SA-ER and SA-IR)
  * Part IV: 6 g/day or 12 g/day SA (SA-ER only)
Arm/Group | Crossover Participants; 6 g/Day | Crossover Participants: 12 g/Day | Crossover Participants: Any Dose | Naïve Participants: 6 g/Day | Naïve Participants: 12 g/Day | Overall: Any Dose
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46 | 0/46 | 0/1 | 0/13 | 0/59
Serious Adverse Events (participants affected / at risk) | 2/46 | 0/46 | 2/46 | 0/1 | 1/13 | 3/59
Other Adverse Events (participants affected / at risk) | 42/46 | 44/46 | 46/46 | 1/1 | 13/13 | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Participants; 6 g/Day (N=46) | Crossover Participants: 12 g/Day (N=46) | Crossover Participants: Any Dose (N=46) | Naïve Participants: 6 g/Day (N=1) | Naïve Participants: 12 g/Day (N=13) | Overall: Any Dose (N=59)
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 — SAE was unrelated to UX001 treatment.
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 — SAE was unrelated to UX001 treatment.
Quadriparesis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 — SAE was unrelated to UX001 treatment.
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1 — SAE was unrelated to UX001 treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Participants; 6 g/Day (N=46) | Crossover Participants: 12 g/Day (N=46) | Crossover Participants: Any Dose (N=46) | Naïve Participants: 6 g/Day (N=1) | Naïve Participants: 12 g/Day (N=13) | Overall: Any Dose (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 0 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 3 | 0 | 3 | 6
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 4 | 0 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 3 | 3 | 5 | 0 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 6 | 0 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 4
Dental caries (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 11 | 13 | 1 | 5 | 18
Dyspepsia (Gastrointestinal disorders) | 3 | 13 | 14 | 0 | 3 | 17
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 8 | 24 | 27 | 0 | 11 | 38
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 2 | 4
Nausea (Gastrointestinal disorders) | 1 | 8 | 8 | 0 | 1 | 9
Toothache (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 2 | 5
Vomiting (Gastrointestinal disorders) | 3 | 4 | 6 | 0 | 1 | 7
Asthenia (General disorders) | 2 | 2 | 3 | 0 | 0 | 3
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 4 | 7 | 1 | 3 | 11
Influenza like illness (General disorders) | 9 | 13 | 17 | 0 | 6 | 23
Malaise (General disorders) | 0 | 1 | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 1 | 3 | 0 | 0 | 3
Pain (General disorders) | 1 | 6 | 7 | 0 | 0 | 7
Peripheral swelling (General disorders) | 2 | 3 | 5 | 1 | 1 | 6
Product taste abnormal (General disorders) | 3 | 0 | 3 | 0 | 0 | 3
Pyrexia (General disorders) | 2 | 6 | 8 | 0 | 1 | 9
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | 3
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 2
Gingivitis (Infections and infestations) | 1 | 2 | 2 | 0 | 1 | 3
Influenza (Infections and infestations) | 1 | 2 | 2 | 0 | 3 | 5
Nasopharyngitis (Infections and infestations) | 3 | 4 | 5 | 0 | 3 | 8
Onychomycosis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 3
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 3 | 6 | 0 | 2 | 8
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 4
Sinusitis (Infections and infestations) | 3 | 4 | 6 | 0 | 1 | 7
Tinea pedis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 2
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4 | 1 | 1 | 6
Urinary tract infection (Infections and infestations) | 1 | 4 | 5 | 0 | 0 | 5
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 8 | 10 | 0 | 5 | 15
Fall (Injury, poisoning and procedural complications) | 4 | 5 | 8 | 0 | 3 | 11
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 4 | 5 | 0 | 2 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0 | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 25 | 0 | 25 | 0 | 2 | 27
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 0 | 3 | 7
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Lipase increased (Investigations) | 3 | 0 | 3 | 0 | 0 | 3
Liver function test abnormal (Investigations) | 3 | 0 | 3 | 0 | 1 | 4
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0 | 0 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 3 | 5 | 0 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 10 | 17 | 0 | 8 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 12 | 17 | 0 | 3 | 20
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0 | 0 | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 0 | 0 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8 | 0 | 1 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 10 | 12 | 0 | 1 | 13
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 1 | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7 | 0 | 2 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 8 | 13 | 1 | 7 | 20
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Decreased vibratory sense (Nervous system disorders) | 2 | 2 | 3 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 5 | 8 | 11 | 0 | 2 | 13
Headache (Nervous system disorders) | 11 | 16 | 21 | 0 | 6 | 27
Hyporeflexia (Nervous system disorders) | 1 | 2 | 3 | 0 | 1 | 4
Migraine (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 3
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 2 | 4 | 0 | 0 | 4
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 3 | 2 | 5 | 0 | 2 | 7
Depression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 0 | 3 | 0 | 1 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1 | 3 | 0 | 1 | 4
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 15 | 0 | 1 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7 | 0 | 2 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 10 | 0 | 5 | 15
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7 | 0 | 0 | 7
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 3
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 4 | 1 | 5 | 0 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0 | 0 | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 6 | 0 | 1 | 7
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 1 | 2 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT01830972/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT01830972/SAP_001.pdf